CLINICAL TRIAL: NCT01291992
Title: Seizures After Cardiac Surgery -- A Prospective Study With Continuous EEG Monitoring
Brief Title: Seizures After Cardiac Surgery -- A Study With Continuous EEG Monitoring
Status: Completed | Type: Observational
Sponsor: London Health Sciences Centre Research Institute OR Lawson Research Institute of St. Joseph's (Other)
Responsible Party: Principal Investigator, Michael Chu, Dr. Michael Chu, London Health Sciences Centre Research Institute OR Lawson Research Institute of St. Joseph's
Other Study IDs: R-10-259; 17107 (Other: REB)
Record Dates: First submitted 2011-02-07; First posted 2011-02-09 (Estimated); Last update posted 2018-03-13 (Actual); Status verified 2018-03

CONDITIONS: Non-convulsive Seizures
Keywords: Non-convulsive seizures; Cardiac Surgery; Postop; 24 hour EEG Monitoring

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Continuous EEG Monitoring: Immediately after surgery, while still sedated and in the cardiac surgery recovery unit, 9 sticker electrodes applied to the skin just below the hairline, which record brain activity onto a computer. The EEG will be recorded for 24 hours. This brain activity (EEG) will later be interpreted by a neurologist who will be looking for evidence of seizure activity in the brain waves. Other relevant information: age, sex, the nature of other health problems, drugs used, complications and whether or not seizures are found will be stored on our computer for further evaluation.

SUMMARY:
The aim of this study is to determine the frequency of nonconvulsive seizures after cardiac surgery using an electroencephalogram or EEG, which records brainwaves through the scalp.

DETAILED DESCRIPTION:
Background: Most patients do not have any neurological complications after cardiac surgery, but fewer than 1% may have a seizure (abnormal brain activity), with or without a convulsion. This can be due to a reaction to certain types of drugs or less commonly stroke or inflammation. Some seizures in post-operative and intensive care unit patients do not result in convulsions, but rather the abnormal brain activity simply causes confusion or unresponsiveness. The incidence of this type of "nonconvulsive"seizure after cardiac surgery is unknown.

Purpose of the study: The aim of this study is to determine the frequency of nonconvulsive seizures after cardiac surgery using an electroencephalogram or EEG, which records brainwaves through the scalp.

Design of the study: The investigators target is to enroll 150 patients undergoing cardiac surgery. The investigators are including patients greater than 18 years of age who are admitted to the CSRU immediately after cardiac surgery. Included patients are of normal mentation and are able to give their own consent. The investigators will exclude only those patients for whom technical issues prevent us from recording the EEG.

ELIGIBILITY:
Inclusion Criteria:

* All adult patients able to give informed consent and undergoing cardiac surgery

Exclusion Criteria:

* Inability to record subhairline EEG data due to technical/mechanical reasons Patients not giving informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All patients admitted to the CSRU postoperatively who have given informed consent to have immediate and continous EEG monitoring for the first 24 hours postoperatively
Sampling Method: Non-Probability Sample
Enrollment: 100 (Actual)
Dates: Start 2010-09 (Actual); Primary Completion 2012-10 (Actual); Study Completion 2013-01 (Actual)

PRIMARY OUTCOMES:
Frequency of non-convulsive seizures in postoperative cardiac surgery patients | Immediate postoperative monitoring with continuous EEG
  Immediately after surgery, while still sedated and in the cardiac surgery recovery unit, 9 sticker electrodes will be applied to the skin just below the hairline, which record brain activity onto a computer. The EEG will be recorded for 24 hours. This brain activity (EEG) will later be interpreted by a neurologist who will be looking for evidence of seizure activity in the brain waves. Other relevant information: age, sex, the nature of other health problems, drugs used, complications and whether or not seizures are found will be stored on our computer for further evaluation.

CONTACTS AND LOCATIONS:
Overall Officials: Michael Chu, MD, Principal Investigator — London Health Sciences Centre, University Hospital
Locations (1):
- London Health Sciences Centre, University Hospital, London, Ontario, Canada

REFERENCES:
- [Background] Bucerius J, Gummert JF, Borger MA, Walther T, Doll N, Onnasch JF, Metz S, Falk V, Mohr FW. Stroke after cardiac surgery: a risk factor analysis of 16,184 consecutive adult patients. Ann Thorac Surg. 2003 Feb;75(2):472-8. doi: 10.1016/s0003-4975(02)04370-9. PMID 12607656
- [Background] Roach GW, Kanchuger M, Mangano CM, Newman M, Nussmeier N, Wolman R, Aggarwal A, Marschall K, Graham SH, Ley C. Adverse cerebral outcomes after coronary bypass surgery. Multicenter Study of Perioperative Ischemia Research Group and the Ischemia Research and Education Foundation Investigators. N Engl J Med. 1996 Dec 19;335(25):1857-63. doi: 10.1056/NEJM199612193352501. PMID 8948560
- [Background] Young GB, Jordan KG, Doig GS. An assessment of nonconvulsive seizures in the intensive care unit using continuous EEG monitoring: an investigation of variables associated with mortality. Neurology. 1996 Jul;47(1):83-9. doi: 10.1212/wnl.47.1.83. PMID 8710130
- [Background] Jordan KG. Continuous EEG and evoked potential monitoring in the neuroscience intensive care unit. J Clin Neurophysiol. 1993 Oct;10(4):445-75. doi: 10.1097/00004691-199310000-00006. PMID 8308143
- [Background] Furtmuller R, Schlag MG, Berger M, Hopf R, Huck S, Sieghart W, Redl H. Tranexamic acid, a widely used antifibrinolytic agent, causes convulsions by a gamma-aminobutyric acid(A) receptor antagonistic effect. J Pharmacol Exp Ther. 2002 Apr;301(1):168-73. doi: 10.1124/jpet.301.1.168. PMID 11907171
- [Background] Mohseni K, Jafari A, Nobahar MR, Arami A. Polymyoclonus seizure resulting from accidental injection of tranexamic acid in spinal anesthesia. Anesth Analg. 2009 Jun;108(6):1984-6. doi: 10.1213/ane.0b013e3181a04d69. PMID 19448237
- [Background] Murkin JM, Falter F, Granton J, Young B, Burt C, Chu M. High-dose tranexamic Acid is associated with nonischemic clinical seizures in cardiac surgical patients. Anesth Analg. 2010 Feb 1;110(2):350-3. doi: 10.1213/ANE.0b013e3181c92b23. Epub 2009 Dec 8. PMID 19996135
- [Derived] Gofton TE, Chu MW, Norton L, Fox SA, Chase L, Murkin JM, Young GB. A prospective observational study of seizures after cardiac surgery using continuous EEG monitoring. Neurocrit Care. 2014 Oct;21(2):220-7. doi: 10.1007/s12028-014-9967-x. PMID 24710654